CLINICAL TRIAL: NCT03760302
Title: Analgesia in ÖAMTC Helicopter Emergency Service in Austria: A Retrospective Analysis
Brief Title: Analgesia in ÖAMTC Helicopter Emergency Service in Austria
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: AN2015-0068 347/4.13 381/5.19
Record Dates: First submitted 2018-11-26; First posted 2018-11-30 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Field Physician Care; Analgesics; Hypnotics; Emergencies; Safety; Accident; Trauma, Multiple; Pain, Acute
MeSH Terms: conditions — Emergencies; Multiple Trauma; Acute Pain | interventions — Analgesics; Hypnotics and Sedatives

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient given analgesics or hypnotics: All patients treated with any kind of analgesics or hypnotics are analyzed and compared.
  Interventions: Other: analgesics; Other: hypnotics

INTERVENTIONS:
Other: analgesics — analgesics given to a patient treated from HEMS
Other: hypnotics — hypnotics given to a patient treated from HEMS

SUMMARY:
A sufficient analgesia in injured or sick people is the main goal of physicians treating a patient. In emergency medicine potent analgesia like ketamine or opioids are routinely used. It is unknown if there are any severe side effects or if the use is safe while in use in a Helicopter Emergency Service equipped with emergency physicians.

ELIGIBILITY:
Inclusion Criteria:

* Analgesia or use of hypnotics in ÖAMTC Air Ambulance Service in Austria 2000-2016

Exclusion Criteria:

* No analgesia, or analgesia use not in connection to ÖAMTC Air Ambulance Service. Analgesia given not in the period of examination (2000-2016)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients screened with the described inclusion criteria - eligible to be included in analysis.
Sampling Method: Probability Sample
Enrollment: 35000 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-10-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Successful analgesia | 2000-2016
  Change in reported pain severity before and after treatment with analgesic. (Numeric Rating Scale, NRS, eleven-point scale reporting no pain=0, to maximum pain=10; 1-3 mild pain, 4-6 moderate pain, 7-10 severe pain)
Analgesic, drug type | 2000-2016
  Use of analgesic (n= type of analgesic)
Analgesic, frequency | 2000-2016
  Use of analgesic (n= frequency how often analgesic is used)
Analgesic, amount of analgesics | 2000-2016
  Use of analgesic (n= amount of analgesic used in mg or µg)

SECONDARY OUTCOMES:
Side effects | 2000-2016
  Type of side effect (respiratory arrest after use, hypoxemia, desaturation (SpO2<90%), dead)
Frequency of side effects | 2000-2016
  Frequency of side effects (frequency of side effect/n=total number of analgesic use; very common>=1/10, common>=1/100 and<1/10, uncommon >=1/1000 and <1/100, rare >=1/10000 and <1/1000, very rare <1/10000)
Severity of side effect | 2000-2016
  severity of side effect (0=none, 1=mild, 2=moderate, 3=severe, 4=potentially life threatening)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ströhle, Dr, Principal Investigator — General and Surgical Critical Care Medicine, Medical University of Innsbruck
Locations (1):
- General and Surgical Critical Care Medicine, Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No